CLINICAL TRIAL: NCT04536246
Title: Comparison of Functional Outcome Between Bone Quadriceps Tendon (BQT) and Single-Bundle Hamstring Tendon (SBHT) Autograft in Arthroscopic-assissted Anterior Cruciate Ligament Reconstruction: a Prospective Cohort Study
Brief Title: Comparison of Functional Outcome Between BQT and SBHT ACL Reconstruction
Acronym: BQTSBHTFMUI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Andri Maruli Tua Lubis, Head of Orthopaedic Sports and Arthroscopy Division, Principal Investigator, Indonesia University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BQT-SBHT-FMUI
Record Dates: First submitted 2020-07-16; First posted 2020-09-02 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Sports Injury; Anterior Cruciate Ligament Rupture
Keywords: ACL reconstruction; Arthroscopic-assisted; BQT; SBHT
MeSH Terms: conditions — Athletic Injuries; Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Intervention Model Description: multi-site study 15 subjects on each group analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BQT Group (Active Comparator): Procedure on this arm = bone quadriceps tendon reconstruction
  Interventions: Procedure: Bone Quadriceps Tendon (BQT) arthroscopic-assisted ACL reconstruction
- SBHT Group (Other): Procedure on this arm = single-bundle hamstring tendon reconstruction
  Interventions: Procedure: Single-Bundle Hamstring Tendon (SBHT) arthroscopic-assisted ACL reconstruction

INTERVENTIONS:
Procedure: Bone Quadriceps Tendon (BQT) arthroscopic-assisted ACL reconstruction — New intervention method deployed in Indonesia to gain better clinical outcome for ACL--deficient patients requiring surgical treatment
  Arms: BQT Group
Procedure: Single-Bundle Hamstring Tendon (SBHT) arthroscopic-assisted ACL reconstruction — Comparator for New Reconstruction Technique
  Arms: SBHT Group

SUMMARY:
ACL rupture has a high morbidity in productive-age population. The increasing incidence and proper management has become a point of interest in the musculoskeletal sport injury. Choosing the best graft has become the main focus in searching for a better outcome regarding ACL reconstruction in these patient population. Currently, single bundle hamstring tendon (SBHT) autograft was preferred in Asian population compared to bone quadriceps tendon (BQT) autograft. However, there are some problems such as smaller size, as well as diameter, of SBHT. This study is focused on evaluation of the clinical outcome between BQT and SBHT in arthroscopic-assisted ACL reconstruction patients.

DETAILED DESCRIPTION:
In this prospective cohort study, 30 subjects were divided into 2 groups (BQT and SBHT). Sampling was taken between February 2016-2017 (1 year) in one orthopaedic center. The instruments used for evaluation are rolimeter and PRO questionnaires (IKDC, Tegner-Lysholm, and KOOS) with data mining between 1 month, 3 months, and 6 months post operation.

To obtain a valid and accountable research data, the investigators collected the information based on 2 parameters and then crosschecked the results.

After clinical data was obtained, the investigators translate the results into a statistical data using SPSS ver.24 and simplified the data for national registry and academic purposes.

According to previous studies, and research hypothesis, functional outcome of patient undergoing arthroscopic-assisted ACL reconstruction is better in BQT group compared to SBHT group, both in subjective and objective parameters given.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral, total rupture of ACL
* Procedure performed by the same surgeon
* Age of subjects between 15-40 years old

Exclusion Criteria:

* Multiligamentous injury
* Bilateral ACL ruptures
* Ligamentous laxity
* Prior knee ligamentous surgery

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2017-11-17 (Actual)

PRIMARY OUTCOMES:
Changes (Improvement) of Rolimeter Measurement After Procedure | Measurement in 1 year after operation
  1. Rolimeter measurement is the objective outcome expected in this study
  2. This device was calibrated and tested prior to the usage in the study
  3. Literature review --> no significant difference between KT1000/2000 and rolimeter for measuring antero-posterior translation of the knee joint
Changes (Improvement) of PRO Questionnaire After Procedure | PRO was taken in a period of 1 year after surgical procedure
  1. We use three different PRO to make an accountable subjective outcome
  2. No standard PRO questionnaire for ACL cases; we used three to be able to triangulate the mean subjective outcome
  3. Rationale for using three PRO : these PROs were rapidly used in other similar studies around the world, had good and reliable results, and contains categoric and numeric data for statistical computation and interpretation

REFERENCES:
- [Background] Cavaignac E, Coulin B, Tscholl P, Nik Mohd Fatmy N, Duthon V, Menetrey J. Is Quadriceps Tendon Autograft a Better Choice Than Hamstring Autograft for Anterior Cruciate Ligament Reconstruction? A Comparative Study With a Mean Follow-up of 3.6 Years. Am J Sports Med. 2017 May;45(6):1326-1332. doi: 10.1177/0363546516688665. Epub 2017 Mar 8. PMID 28273424
- [Background] Lee JK, Lee S, Lee MC. Outcomes of Anatomic Anterior Cruciate Ligament Reconstruction: Bone-Quadriceps Tendon Graft Versus Double-Bundle Hamstring Tendon Graft. Am J Sports Med. 2016 Sep;44(9):2323-9. doi: 10.1177/0363546516650666. Epub 2016 Jun 30. PMID 27365373
- [Background] Haner M, Bierke S, Petersen W. Anterior Cruciate Ligament Revision Surgery: Ipsilateral Quadriceps Versus Contralateral Semitendinosus-Gracilis Autografts. Arthroscopy. 2016 Nov;32(11):2308-2317. doi: 10.1016/j.arthro.2016.03.020. Epub 2016 May 18. PMID 27209621
- [Background] Akoto R, Hoeher J. Anterior cruciate ligament (ACL) reconstruction with quadriceps tendon autograft and press-fit fixation using an anteromedial portal technique. BMC Musculoskelet Disord. 2012 Aug 27;13:161. doi: 10.1186/1471-2474-13-161. PMID 22925587
- [Background] Yue B, Varadarajan KM, Ai S, Tang T, Rubash HE, Li G. Differences of knee anthropometry between Chinese and white men and women. J Arthroplasty. 2011 Jan;26(1):124-30. doi: 10.1016/j.arth.2009.11.020. Epub 2010 Feb 9. PMID 20149574
- [Background] Zaffagnini S, Marcacci M, Lo Presti M, Giordano G, Iacono F, Neri MP. Prospective and randomized evaluation of ACL reconstruction with three techniques: a clinical and radiographic evaluation at 5 years follow-up. Knee Surg Sports Traumatol Arthrosc. 2006 Nov;14(11):1060-9. doi: 10.1007/s00167-006-0130-x. Epub 2006 Aug 15. PMID 16909301
- [Background] Collins NJ, Misra D, Felson DT, Crossley KM, Roos EM. Measures of knee function: International Knee Documentation Committee (IKDC) Subjective Knee Evaluation Form, Knee Injury and Osteoarthritis Outcome Score (KOOS), Knee Injury and Osteoarthritis Outcome Score Physical Function Short Form (KOOS-PS), Knee Outcome Survey Activities of Daily Living Scale (KOS-ADL), Lysholm Knee Scoring Scale, Oxford Knee Score (OKS), Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), Activity Rating Scale (ARS), and Tegner Activity Score (TAS). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11(0 11):S208-28. doi: 10.1002/acr.20632. No abstract available. PMID 22588746
- [Background] Bekkers JE, de Windt TS, Raijmakers NJ, Dhert WJ, Saris DB. Validation of the Knee Injury and Osteoarthritis Outcome Score (KOOS) for the treatment of focal cartilage lesions. Osteoarthritis Cartilage. 2009 Nov;17(11):1434-9. doi: 10.1016/j.joca.2009.04.019. Epub 2009 May 7. PMID 19454278
- [Background] Schulz AP, Lange V, Gille J, Voigt C, Frohlich S, Stuhr M, Jurgens C. Anterior cruciate ligament reconstruction using bone plug-free quadriceps tendon autograft: intermediate-term clinical outcome after 24-36 months. Open Access J Sports Med. 2013 Nov 19;4:243-9. doi: 10.2147/OAJSM.S49223. eCollection 2013. PMID 24379730
- [Background] Mologne T, Friedman M. Arthroscopic anterior cruciate reconstruction with hamstring tendons: indications, surgical technique, and complications and their treatment. In: Insall & Scott Surgery of the Knee. 4th ed. Philadelphia: Elsevier Inc; 2006.
- [Background] Chen V, Hunter R, Woolf J. Anterior Cruciate Ligament Injuries. In: Schepsis A, Busconi B, editors. Orthopaedic Surgery Essential - Sports Medicine. Philadelphia: Lippincott Williams & Wilkins; 2006.
- [Background] Pavlovich R Jr, Goldberg SH, Bach BR Jr. Adolescent ACL injury: treatment considerations. J Knee Surg. 2004 Apr;17(2):79-93. doi: 10.1055/s-0030-1248203. PMID 15124660
- [Background] Lyman S, Koulouvaris P, Sherman S, Do H, Mandl LA, Marx RG. Epidemiology of anterior cruciate ligament reconstruction: trends, readmissions, and subsequent knee surgery. J Bone Joint Surg Am. 2009 Oct;91(10):2321-8. doi: 10.2106/JBJS.H.00539. PMID 19797565
- [Background] Shi DL, Yao ZJ. Knee function after anterior cruciate ligament reconstruction with patellar or hamstring tendon: a meta-analysis. Chin Med J (Engl). 2011 Dec;124(23):4056-62. PMID 22340342
- [Background] Peter Layde SLC, Layde P, Guse CE, Schlotthauer AE, Valin SE Van. The Incidence and Etiology of Anterior Cruciate Ligament Injuries in Patients under the Age of 18 in the State of Wisconsin. Pediatr Ther [Internet]. 2014;04(02). Available from: https://www.omicsonline.org/open-access/the-incidence-and-etiology-of-anterior-cruciate-ligament-injuries-in-patients-under-the-age-of-in-the-state-of-wisconsin-2161-0665.1000196.php?aid=26065
- [Background] Collins JE, Katz JN, Donnell-Fink LA, Martin SD, Losina E. Cumulative incidence of ACL reconstruction after ACL injury in adults: role of age, sex, and race. Am J Sports Med. 2013 Mar;41(3):544-9. doi: 10.1177/0363546512472042. Epub 2013 Jan 9. PMID 23302260
- [Background] Tow BP, Chang PC, Mitra AK, Tay BK, Wong MC. Comparing 2-year outcomes of anterior cruciate ligament reconstruction using either patella-tendon or semitendinosus-tendon autografts: a non-randomised prospective study. J Orthop Surg (Hong Kong). 2005 Aug;13(2):139-46. doi: 10.1177/230949900501300206. PMID 16131675
- [Background] Deehan DJ, Salmon LJ, Webb VJ, Davies A, Pinczewski LA. Endoscopic reconstruction of the anterior cruciate ligament with an ipsilateral patellar tendon autograft. A prospective longitudinal five-year study. J Bone Joint Surg Br. 2000 Sep;82(7):984-91. doi: 10.1302/0301-620x.82b7.10573. PMID 11041586
- [Background] Panni AS, Milano G, Tartarone M, Demontis A, Fabbriciani C. Clinical and radiographic results of ACL reconstruction: a 5- to 7-year follow-up study of outside-in versus inside-out reconstruction techniques. Knee Surg Sports Traumatol Arthrosc. 2001;9(2):77-85. doi: 10.1007/s001670000171. PMID 11354857
- [Background] Dargel J, Schmidt-Wiethoff R, Schneider T, Bruggemann GP, Koebke J. Biomechanical testing of quadriceps tendon-patellar bone grafts: an alternative graft source for press-fit anterior cruciate ligament reconstruction? Arch Orthop Trauma Surg. 2006 May;126(4):265-70. doi: 10.1007/s00402-005-0048-7. Epub 2005 Sep 17. PMID 16172862
- [Background] Staeubli HU, Bollmann C, Kreutz R, Becker W, Rauschning W. Quantification of intact quadriceps tendon, quadriceps tendon insertion, and suprapatellar fat pad: MR arthrography, anatomy, and cryosections in the sagittal plane. AJR Am J Roentgenol. 1999 Sep;173(3):691-8. doi: 10.2214/ajr.173.3.10470905.
- [Background] Lee S, Seong SC, Jo H, Park YK, Lee MC. Outcome of anterior cruciate ligament reconstruction using quadriceps tendon autograft. Arthroscopy. 2004 Oct;20(8):795-802. doi: 10.1016/j.arthro.2004.06.009. PMID 15483539
- [Background] Beynnon BD, Johnson RJ, Abate JA, Fleming BC, Nichols CE. Treatment of anterior cruciate ligament injuries, part 2. Am J Sports Med. 2005 Nov;33(11):1751-67. doi: 10.1177/0363546505279922. PMID 16230470
- [Background] Sofu H, Sahin V, Gursu S, Yildirim T, Issin A, Ordueri M. Use of quadriceps tendon versus hamstring tendon autograft for arthroscopic anterior cruciate ligament reconstruction: a comparative analysis of clinical results. Eklem Hastalik Cerrahisi. 2013;24(3):139-43. doi: 10.5606/ehc.2013.31. PMID 24191878
- [Background] van Eck CF, Kropf EJ, Romanowski JR, Lesniak BP, Tranovich MJ, van Dijk CN, Fu FH. Factors that influence the intra-articular rupture pattern of the ACL graft following single-bundle reconstruction. Knee Surg Sports Traumatol Arthrosc. 2011 Aug;19(8):1243-8. doi: 10.1007/s00167-011-1427-y. Epub 2011 Feb 11. PMID 21311861
- [Background] Ramski DE, Kanj WW, Franklin CC, Baldwin KD, Ganley TJ. Anterior cruciate ligament tears in children and adolescents: a meta-analysis of nonoperative versus operative treatment. Am J Sports Med. 2014 Nov;42(11):2769-76. doi: 10.1177/0363546513510889. Epub 2013 Dec 4. PMID 24305648